CLINICAL TRIAL: NCT02020265
Title: Longitudinal Study of the Effect of Neurofeedback Training on Soldiers Emotional Regulation Ability and Mental Resilience to Stress.
Brief Title: fMRI Based EEG Neurofeedback as a Method of Enhancing Emotional Resilience Among Soldiers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0080-13
Record Dates: First submitted 2013-11-12; First posted 2013-12-24 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Stress; Depression
Keywords: stress and depression related symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- NF group (Experimental): This group will train modulation of the amygdala EEG fingerprint by EEG neurofeedback.
  Interventions: Device: EEG neurofeedback
- Sham NF (Sham Comparator): This group preform the same procedure as the NF group only reviving sham feedback
  Interventions: Device: EEG neurofeedback
- A\T NF (Active Comparator): This group will train modulation of A\T ratio by EEG neurofeedback
  Interventions: Device: EEG neurofeedback

INTERVENTIONS:
Device: EEG neurofeedback

SUMMARY:
EEG protocols exist for reducing stress and improve PTSD symptoms (A/T EEG protocols, Peniston, 1993, Hammond, 2005) however; our innovative EEG-NF LMI approach intends to be more amygdala/stress specific and therefore more efficient. Three groups of soldiers, while in operational activity will go through 24 sessions of 3 different methods of EEG-NF; our newly developed NF via MLI, a standard procedure for NF via A/T and a placebo NF. Difference between the groups in regard to their emotion regulation capability will be tested by fMRI with regard to amygdala activation following EEG-NF LMI as well as two stress challenge tests.

ELIGIBILITY:
Inclusion Criteria:

* soldiers in preliminary combat training

Exclusion Criteria:

* known mental disorders or neuro-pathology

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-02; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline at Amygdala modulation ability | At baseline and after 6 month of neurofeeback training.
  The test group will show a grater improvment from baseline in amygdala modulation abilities as measured by real time fMRI

SECONDARY OUTCOMES:
Change from baseline in Emotion regulation ability | At baseline and after 6 month of neurofeedback training
  The test group will show grater improvement from baseline of emotion regulation abilities as measured by implicit and explicit test and by fMRI

CONTACTS AND LOCATIONS:
Locations (1):
- Tel-Aviv Sourasky medical center, Tel_Aviv, Choose One, Israel